CLINICAL TRIAL: NCT00819611
Title: Working Memory Training: A Randomised Controlled Treatment Study in Young ADHD Children
Brief Title: Working Memory Training in Young ADHD Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Netherlands Organisation for Scientific Research (Other Government)
Responsible Party: Principal Investigator, Dorine Slaats, PhD, Radboud University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WM01022009; RN000142
Record Dates: First submitted 2009-01-08; First posted 2009-01-09 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2014-01

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: Attention deficit disorder with hyperactivity; Working memory training; Placebo; Behavioral symptoms; Neuropsychology; Electropsychophysiology
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Behavioral Symptoms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Working memory training (Experimental)
  Interventions: Behavioral: Cogmed Working memory training
- Control version of working memory training (Sham Comparator)
  Interventions: Behavioral: Control version of Cogmed working memory training

INTERVENTIONS:
Behavioral: Cogmed Working memory training — 15 minutes of working memory training, 5 days a week for a period of 5 weeks
  Arms: Working memory training
Behavioral: Control version of Cogmed working memory training — 15 minutes of 'sham' working memory training, 5 days a week for a period of 5 weeks
  Arms: Control version of working memory training

SUMMARY:
The purpose of this study is to investigate whether working memory training improves behavioral symptoms, neurocognitive performance, and neural functioning in young children with ADHD.

ELIGIBILITY:
Inclusion Criteria:

* Age between 4 years/6 months and 7 years/4 months
* Diagnosis ADHD, classified by the DSM-IV (Diagnostic and Statistical Manual of Mental Disorders, 2000)
* A full scale IQ >= 80
* Psychopharmaca- naïve or -free
* Access to a PC with Windows Vista or Windows XP with internet connection and speakers at home

Exclusion Criteria:

* Currently intensive (i.e. weekly) individual or group psychotherapy
* Regular use of medication
* Diagnosis of one or more of the following comorbid psychiatric disorders: Major depression, Bipolar disorder, Psychotic disorder, Chronically motor tic disorder or Gilles de la Tourette, Conduct disorder, any other autism spectrum disorder except for Pervasive Developmental Disorder Not Otherwise Specified (PDD-NOS), Eating disorders, Anxiety disorders
* Neurological disorders (e.g. epilepsy) currently or in the past
* Cardiovascular disease currently or in the past
* Serious motor or perceptual handicap
* Participation in another clinical trial simultaneously
* Educational level and/ or socio-economic situation that makes it unlikely for the family to fulfil this study

Ages: 54 Months to 88 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2009-06; Primary Completion 2013-05 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
ADHD criteria according to the DSM-IV-TR rated by the investigator | 7 weeks

SECONDARY OUTCOMES:
Neurocognitive performance and electrocortical activity | 7 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dorine Slaats-Willemse, PhD, Principal Investigator — Karakter University Centre for Child and Adolescent Psychiatry, Nijmegen
Locations (1):
- Karakter University Centre for Child and Adolescent Psychiatry Nijmegen, Nijmegen, Netherlands

REFERENCES:
- [Background] Klingberg T, Fernell E, Olesen PJ, Johnson M, Gustafsson P, Dahlstrom K, Gillberg CG, Forssberg H, Westerberg H. Computerized training of working memory in children with ADHD--a randomized, controlled trial. J Am Acad Child Adolesc Psychiatry. 2005 Feb;44(2):177-86. doi: 10.1097/00004583-200502000-00010. PMID 15689731
- [Derived] van Dongen-Boomsma M, Vollebregt MA, Buitelaar JK, Slaats-Willemse D. Working memory training in young children with ADHD: a randomized placebo-controlled trial. J Child Psychol Psychiatry. 2014 Aug;55(8):886-96. doi: 10.1111/jcpp.12218. Epub 2014 Mar 15. PMID 24628438